CLINICAL TRIAL: NCT01423617
Title: Double-blind, Randomized, Placebo-controlled, Bicentric Study to Evaluate the Safety and Efficacy of Zenoctil in Reducing Body Weight of Overweight Subjects
Brief Title: Efficacy and Safety of Zenoctil in Reducing Body Weight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INQ/005611
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Overweight
Keywords: overweight; weight loss; body fat; waist circumference; satiety; appetite
MeSH Terms: conditions — Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zenoctil (Active Comparator)
  Interventions: Dietary Supplement: Zenoctil
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Zenoctil — 3 tablets 2 times daily
  Arms: Zenoctil
Other: Placebo — 3 tablets 2 times daily
  Arms: Placebo

SUMMARY:
The intention of the study is to evaluate the safety and potential body weight and body fat loss effects of a 12-week treatment with Zenoctil in a randomized, double-blind, placebo-controlled, parallel study conducted in Caucasian subjects.

This study will also include a diet plan for each subject, calculated based on gender, age, and energy requirements; and adjusted to be slightly hypocaloric.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian males and females, age 18 to 60 years
* 25 kg/m2 ≤ BMI ≤32 kg/m2
* Expressed desire for weight loss
* Accustomed to 3 main meals a day
* Consistent and stable body weight 3 months prior to study enrollment
* Commitment to avoid the use of other weight loss products/programs during the study
* Commitment to adhere to diet recommendation
* Females' agreement to use appropriate birth control methods during the active study period
* Subject declares in writing his/her consent to participate, understands requirements of the study and is willing to comply

Exclusion Criteria:

* Known sensitivity to Garcinia cambogia, Lagerstroemia speciosa (other members of Lythraceae family), caffeine, tannins
* History of diabetes mellitus or other endocrine disorders
* Fasting blood glucose >7 mmol/L
* Treatment with systemic corticosteroids within the last 12 months
* Current use of antidepressants
* Uncontrolled hypertension (>160/110) or other uncontrolled cardiac, pulmonary, renal, or liver disease, determined to be clinically significant by the investigator
* Presence of acute or history of chronic gastrointestinal disease
* Schizophrenia or other diagnosed psychiatric disorders
* Any other acute or chronic disease or any other medical condition which, in the investigator's view, may preclude subject's inclusion (e.g., cancer, HIV)
* Bariatric surgery
* Abdominal surgery within the last 6 months
* History of eating disorders like bulimia, anorexia nervosa
* Changes in the dose of estrogen, contraceptives or thyroid hormone within the last 3 months
* Pregnancy or nursing
* Any medication or use of products for the treatment of obesity (e.g., fat binder, carbohydrate blocker/starch blocker, fat burner, satiety products etc.) within the last 6 weeks
* More than 3 hours strenuous sport activity per week
* History of abuse of drugs, alcohol or medication
* Smoking cessation within the 6 months prior to this study
* Incompliance due to language difficulties
* Participation in another study during the last 4 weeks
* Clinically relevant excursions of safety parameters

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Grube, MD, Principal Investigator
Locations (1):
- Barbara Grube, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zenoctil | Placebo
Started | 46 | 46
Completed | 46 | 45
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zenoctil | Placebo | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (10.9) | 42.5 (11.6) | 42.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 62
  Male | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Body Weight (kg)
Description: Change in mean body weight at week 12 compared to baseline.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Zenoctil | Placebo
Number analyzed (Participants) | 46 | 45
kg | -2.26 (2.37) | -0.56 (2.45)

2. Primary Outcome: Change in Mean Body Fat (kg)
Description: Change in mean body fat at week 12 compared to baseline
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Zenoctil | Placebo
Number analyzed (Participants) | 46 | 45
kg | -1.12 (1.84) | 0.37 (2.14)

3. Secondary Outcome: Number of Subjects Who Lost at Least 3% of Baseline Body Weight
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Zenoctil | Placebo
Number analyzed (Participants) | 46 | 45
participants | 24 | 8

4. Secondary Outcome: Changes in Waist Circumference (cm)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Zenoctil | Placebo
Number analyzed (Participants) | 46 | 45
cm | -2.00 (2.44) | -0.69 (2.24)

5. Secondary Outcome: Changes in Hip Circumference
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Zenoctil | Placebo
Number analyzed (Participants) | 46 | 45
cm | -1.54 (1.76) | 0.64 (1.91)

6. Secondary Outcome: Changes in Waist-hip-ratio
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Changes in Body Fat Content (%)
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Changes in Hunger, Eating, and Food-craving Related Items From the Control of Eating Questionnaire (COEQ)
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Subjects' Global Feeling of Satiety
Description: Subject's feeling of satiety (subsequent to the three main meals) is judged globally by the subjects on the basis of a 4 point rating scale: 0 = "no"; 1 = "slightly", 2 = "moderate" and 3 = "strong".
Time Frame: 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Changes in Body Fat Free Mass (kg)
Time Frame: 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Global Evaluation of Safety by Investigators
Description: The investigators evaluate independently the safety of the investigational product, using a scale with scores of "very good", "good", "moderate" and "poor".
Time Frame: 12 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Global Evaluation of Safety by Subjects
Description: The subjects evaluate independently the safety of the investigational product, using a scale with scores of "very good", "good", "moderate" and "poor".
Time Frame: 12 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Global Evaluation of Efficacy by Subjects
Description: The subjects evaluate independently the efficacy of the investigational product, using a scale with scores of "very good", "good", "moderate" and "poor".
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Zenoctil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other